CLINICAL TRIAL: NCT02419690
Title: Effectiveness of a Patient Centered Intervention to Increase Dual Protection Against Unintended Pregnancy and Sexually Transmitted Disease Among Adolescents
Brief Title: Sexual Health Texting Intervention to Support Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Deborah Rinehart, Associate Research Scientist, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-3219
Record Dates: First submitted 2015-01-13; First posted 2015-04-17 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-09

CONDITIONS: Teen Sexual Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The current standard of care in the clinic is a preventive care physical examination every 1-2 years and/or treatment for presenting medical conditions. The frequency and content of reproductive health is not standardized between clinicians, but it is expected that all clinicians will address sexuality during routine visits. Additionally, sexually active teens are encouraged to have urine screening tests for chlamydia, gonorrhea and pregnancy as indicated. Teens may also see a reproductive health educator at the clinic as well. Available contraceptive methods are oral contraceptive pills, contraceptive patches, Depo-Provera, diaphragms, condoms, implants and intrauterine devices (IUDs).
- text message intervention (Active Comparator): Subjects in the intervention arm will receive usual care plus text messages that have been developed to promote overall teen sexual health.
  Interventions: Behavioral: text message intervention

INTERVENTIONS:
Behavioral: text message intervention — Subjects will be sent 58 messages (3-5 per week) over 12 weeks, plus reminder messages for follow up interviews. The content of these messages will focus on contraception methods and effectiveness, sexually transmitted infection (STI) transmission, condom use, partner and parental communication, and healthy relationships. There will also be several text messages asking the participant if they would like to have a health educator contact them. The format will include facts, quizzes, true/false and some will have links to videos/pictures and websites, and some will request a response.
  Arms: text message intervention

SUMMARY:
This study aims to use a text messaging intervention to prevent unintended teen pregnancy and transmission of sexually transmitted disease. The study will be informed by a formative qualitative phase (February 2014 - January 2015) which will include individual qualitative interviews and focus groups with teens to elucidate and explore the barriers to effective contraceptive use and sexually transmitted disease (STD) prevention and to obtain feedback on the developed intervention. The second efficacy phase will randomize subjects to the texting intervention or to usual care.

DETAILED DESCRIPTION:
Adolescents, particularly those from disadvantaged backgrounds, are disproportionally affected by both unintended pregnancies and STDs. While youth only represent a quarter of the sexually active population in the US, they account for almost half of all new STDs and the rate of unintended pregnancies among sexually active teens is almost double the rate of all sexually active women. Teen mothers experience higher rates of negative social outcomes including school dropout and children of teens are more likely to have low birth weight, lower academic achievement and more likely to perpetuate the cycle of teen pregnancy themselves. Both unintended pregnancies and STDs are much higher among racial/ethnic minority populations. Contraceptive methods considered most effective for pregnancy prevention do not protect against STDs and HIV transmission. Dual protection methods include being on an effective and consistent form of contraception and having an effective STD prevention method in place, preferably consistent condom use. Non-penetrative sexual practices can be substituted.

There are many barriers to providing sexual health education and services in the context of primary care visits. A recent study of pediatricians found that 61% of pediatricians reported discussing contraception, use of condoms and/or STDs with patients at preventive care visits. Most providers (76%), however, believed they did not have sufficient time to provide such counseling in the visit. The problems are even more acute in resource-limited safety net settings. Therefore, a two-tiered approach may prove to be useful, where providers initially address reproductive health issues in the visit but where additional support outside the visit provides additional information, support, motivation and connection to services. An innovative intervention using texting technology may prove to be a cost effective method of providing support between visits.

ELIGIBILITY:
Inclusion Criteria:

* biologically female;
* between 13 and 18 years of age;
* not currently pregnant or trying to become pregnant;
* have texting capability; and
* able to read/write/speak in English.

Exclusion Criteria:

* not meeting inclusion criteria outlined above

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 244 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Rinehart, PhD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Text Message Intervention
Started | 122 | 122
Completed | 122 | 122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Text Message Intervention | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 122 | 122 | 244
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (1.7) | 15.7 (1.6) | 15.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 122 | 244
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latinx | 99 | 96 | 195
  White | 14 | 11 | 25
  Black | 8 | 13 | 21
  Asian | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 122 | 122 | 244

OUTCOME MEASURES:

1. Primary Outcome: Dual Protection Behaviors, Reported in Surveys and Reviewed in the Medical Record.
Description: Practice of protection from STIs and unintended pregnancy were reported at baseline and follow up surveys. Between-group differences at baseline, 3 and 6-month follow-up among participants with data at all points AND who were sexually active at baseline were analyzed.
Time Frame: 6 months
Population: For each group, baseline, 3 and 6-month follow-up among participants with data at all points (3 and 6 month follow-up) AND who were sexually active at baseline were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Text Message Intervention
Number analyzed (Participants) | 31 | 33
Participants
  Baseline dual protection behaviors | 7 | 6
  Three-month dual protection behaviors | 8 | 8
  Six-month dual protection behaviors | 7 | 11

2. Secondary Outcome: Use of the Most Effective Contraception Methods: Long Acting Reversible Contraceptives (LARCs)
Description: Use of LARCs was reported at follow up surveys and reviewed in the medical record at 6 months.
Time Frame: 6 months
Population: Between-group differences at baseline, 3 and 6-month follow-up among participants with data at all points. This analysis included those who were not sexually active.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Text Message Intervention
Number analyzed (Participants) | 69 | 67
Participants
  Baseline LARC use | 18 | 16
  Three-month LARC use | 18 | 18
  Six-month LARC use | 17 | 17

3. Secondary Outcome: Knowledge, Motivation, and Attitudes Toward Contraception, Condom Use and Dual Protection in Surveys
Description: Subjects reported their degree of knowledge (0-18, higher score = higher knowledge), motivation (0-12, higher score = higher self-efficacy for condom use), and attitudes (0-40, higher score = more perceived benefits of birth control use) in baseline and follow-up surveys.
Time Frame: 6 months
Population: Between-group differences at baseline, 3 and 6-month follow-up among participants with data at all points were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Text Message Intervention
Number analyzed (Participants) | 69 | 67
score on a scale
  Baseline overall knowledge (0-18) | 10.46 (4.23) | 10.90 (4.03)
  3-month overall knowledge (0-18) | 11.59 (3.94) | 13.57 (3.63)
  6-month overall knowledge (0-18) | 11.97 (4.19) | 13.64 (3.83)
  Baseline self-efficacy condom use (0-12) | 6.97 (1.96) | 7.12 (1.75)
  3-month self-efficacy condom use (0-12) | 6.68 (2.08) | 7.38 (1.76)
  6-month self-efficacy condom use (0-12) | 6.99 (1.82) | 7.39 (1.77)
  Baseline perceived benefits birth control (0-40) | 25.72 (5.40) | 25.90 (5.38)
  3-month perceived benefits birth control (0-40) | 25.59 (5.55) | 27.85 (5.76)
  6-month perceived benefits birth control (0-40) | 26.10 (5.69) | 27.40 (5.59)

4. Secondary Outcome: Unprotected Vaginal Sex at Baseline, 3 and 6 Months Post-baseline (Formerly Incidence of Unintended Pregnancy and STIs)
Description: Urinalysis was to be performed at 6 months post-baseline to test for pregnancy, gonorrhea, and chlamydia. However, the researchers were unable to obtain urinalyses at 6 months from all participants due to logistical challenges and participant attrition. We instead analyzed self-reported unprotected sex (i.e., did not use condoms 100% of the time) at each of the study time points to assess potential risk for unintended pregnancy and/or STI.
Time Frame: 6 months
Population: Between-group differences at baseline, 3 and 6-month follow-up among participants with data at all points AND were sexually active at baseline were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Text Message Intervention
Number analyzed (Participants) | 31 | 33
Participants
  Baseline unprotected vaginal sex | 23 | 26
  3-month unprotected vaginal sex | 18 | 20
  6-month unprotected vaginal sex | 17 | 21

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care | Text Message Intervention
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/122
Other Adverse Events (participants affected / at risk) | 0/122 | 0/122

LIMITATIONS AND CAVEATS:
Data are self-report and thus may be influenced by social desirability and/or recall. Unable to assess 6-month STI and pregnancy incidence. Limited ability to detect significance due to heterogeneous sample and lack of power in stratified analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No